CLINICAL TRIAL: NCT00892398
Title: Trabeculectomy With Mitomycin C Associated With Sub-conjunctival Injection of Ranibizumab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Gisele Li, Assistant Professor, Maisonneuve-Rosemont Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRFB002ACA04T
Record Dates: First submitted 2009-05-01; First posted 2009-05-04 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Glaucoma
Keywords: Trabeculectomy; Vascular Endothelial Growth Factor A; Wound Healing; Angiogenesis Inhibitors
MeSH Terms: conditions — Glaucoma | interventions — Ranibizumab; Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ranibizumab (Experimental): Trabeculectomy with mitomycin C associated with 2 subconjunctival injections of ranibizumab: 1 intraoperatively and 1 at 2 weeks post-operatively
  Interventions: Drug: ranibizumab
- standard care (Active Comparator): Trabeculectomy with mitomycin C and standard post-operative care
  Interventions: Procedure: standard care

INTERVENTIONS:
Drug: ranibizumab — Two ranibizumab subconjunctival injections (0.5 mg ∕ 0.05 mL). The first injection at the end of the surgery (intraoperative) and the second two weeks post-operatively.
  Arms: ranibizumab
Procedure: standard care — standard post-operative care after trabeculectomy with mitomycin C
  Arms: standard care

SUMMARY:
Trabeculectomy with mitomycin C remains the standard surgery for glaucoma. This surgery involves creating a door in the eye wall in order to improve fluid outflow and decrease intraocular pressure. However, success rates range from 70% to 90% depending on the criteria used and tend to decrease with time. The failure of the surgery is associated with inflammation, new blood vessel formation and scarring which can cause closure of the door. Molecules which inhibit new blood vessel formation such as inhibitors of vascular endothelial growth factor have been used successfully to decrease scarring in animal eyes where little doors were created and significantly improve survival. Furthermore, they have shown promise when used during trabeculectomy. Ranibizumab, a vascular endothelial growth factor, has also been used safely in intraocular surgery to treat other diseases which involve new blood vessel formation such as macular degeneration and diabetes.

The investigators hypothesize that ranibizumab may decrease the failure rate of trabeculectomy with mitomycin C by decreasing scarring.

The aim of the study is to evaluate the difference in failure rates and bleb morphology at one year post-operatively in eyes having undergone sub-conjunctival injections of ranibizumab in addition to primary trabeculectomy with mitomycin C compared to eyes having undergone trabeculectomy with mitomycin C alone.

DETAILED DESCRIPTION:
Prospective, randomized, unblinded clinical trial. Two groups of patients with glaucoma undergoing primary trabeculectomy or phaco-trabeculectomy with MMC between March 2009 and September 2012. The ranibizumab group (RAN) received 2 subconjunctival injections of 0.5 mg of ranibizumab (intraoperatively and on day 14) and he control group did not receive ranibizumab.

ELIGIBILITY:
Inclusion Criteria:

* to have uncontrolled glaucoma
* to have accepted to undergo a primary trabeculectomy with mitomycin C
* to have one of the following types of glaucoma:

  * Normal tension Glaucoma
  * Chronic Open-Angle Glaucoma
  * Chronic Angle-Closure Glaucoma
  * Mixed mechanism glaucoma
  * Steroid-induced Glaucoma
  * Neovascular Glaucoma

Exclusion Criteria:

* to be less than 18 years old
* to be unable to observe the study protocol
* to present some risk factors for thromboembolic events and cerebrovascular accidents : hypertension, dyslipidemia, coronary artery diseases
* a history of thromboembolic events and cerebrovascular accidents
* congenital glaucoma
* uveitic glaucoma
* to be pregnant
* to be breastfeeding
* surgical complications prior to injection of the study drug such as vitreous in the anterior chamber or the presence of suprachoroidal hemorrhages
* to have undergone a previous conjunctival surgery
* to be hypersensitive to the drug, to one of the components of the drug or to one of the components of the packaging
* to present an active or suspected intraocular or periocular inflammation
* to have a kidney failure
* to have a liver failure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2009-03; Primary Completion 2013-10 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Failure rates of the surgery as defined by intraocular pressure reductions | one year
  Complete success: post-operative IOP between 5-18 mm Hg and at least a 20% reduction in IOP from baseline without the use of glaucoma medications. Qualified success: similar definition with the use of glaucoma medications.

SECONDARY OUTCOMES:
Bleb morphology using Moorfields bleb grading system | one year

CONTACTS AND LOCATIONS:
Overall Officials: Gisele Li, M.D., Principal Investigator — Maisonneuve-Rosemont Hospital
Locations (1):
- Maisonneuve-Rosemont Hospital, Montreal, Quebec, Canada